CLINICAL TRIAL: NCT06754436
Title: Population Pharmacokinetics of L-AmB in Chinese Patients Assisted by Extracorporeal Membrane Pulmonary Oxygenation (ECMO)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Lin Yang, Director of pharmacy department of Beijing Anzhen Hospital, Beijing Anzhen Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANZHEN HOSPITOL-LY-05
Record Dates: First submitted 2024-12-20; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Invasive Fungal Infections; Liposomal Amphotericin B
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- L-AmB group (Experimental): To establish and validate a population pharmacokinetic model for L-AmB in patients with severe invasive fungal infections treated undergoing ECMO-assisted therapy.
  Interventions: Biological: Determination of blood drug concentration

INTERVENTIONS:
Biological: Determination of blood drug concentration — Collecting blood samples from patients and determining blood drug concentrations. Patients were intravenously titrated after 3 doses of maintenance dose titration of L-AmB. The time points of sample collecting were 30 minutes before and 1, 2, 3, 6, 9, 12, 16, 20, 24 hours after administration. Then, the blood concentrations were determined according to the established method.

SUMMARY:
The goal of this study is to investigate the effects of ECMO-assisted therapy on L-AmB PK parameters in patients with critically ill patients of invasive fungal infections, and to determine the in vivo pharmacokinetic changes of L-AmB in the ECMO population. To establish and validate a population pharmacokinetic model for liposomal amphotericin B in patients with critically ill patients of invasive fungal infections treated with ECMO adjuvant therapy, and to explore the pharmacokinetics/pharmacodynamics of the drug with different dosing regimens.

DETAILED DESCRIPTION:
The information of patient characteristics, physiological parameters, ECMO related parameters, administration and sampling information of L-AmB were collected.Patients were intravenously titrated after 3 doses of maintenance dose titration. The sampling window was from 0 to 24 h. The time points were 0.5 h before and 1, 2, 3, 6, 9, 12, 16, 20 and 24 h after administration. NONMEM software was applied to establish the PPK model of L-AmB.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria for invasive fungal infections presenting to the intensive care unit (ICU) with probable or proved patients According to the 2021 EORTC/MSGERC guideline.
* Requiring ECOM assistance.
* Age 18 years.

Exclusion Criteria:

* Intolerance of L-AmB therapy.
* Pregnancy.
* Expected survival time <24 hours.
* Lack of necessary data on patient demographics physiopathology, and clinical status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2025-11-11 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Blood drug concentration of liposomal amphotericin B | The time points of sample collecting were 30 minutes before and 1, 2, 3, 6, 9, 12, 16, 20, 24 hours after administration.
  Patients were intravenously titrated after 3 doses of maintenance dose titration of L-AmB. Then collecting blood samples from these patients. The blood concentrations of L-AmB were determined according to the established method.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided